CLINICAL TRIAL: NCT02599376
Title: Comparative Study of Haemodynamic Changes After Spinal Anaesthesia in Non-obese and Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1/028/14
Record Dates: First submitted 2014-12-15; First posted 2015-11-06 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Low Cardiac Output
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMI less than 30 (Active Comparator): The drop in cardiac output after spinal anaesthesia for LSCS at various intervals with LiDCORapid
  Interventions: Device: LiDCOrapid
- BMI more than 40 (Experimental): The drop in cardiac output after spinal anaesthesia for LSCS at various intervals with LiDCORapid
  Interventions: Device: LiDCOrapid

INTERVENTIONS:
Device: LiDCOrapid — Cardiac output will be non invasively monitored by using 2 cuffs on fingers.

SUMMARY:
Obesity has become one of the most common risk factors in obstetric practice with serious anaesthetic implications. Obese pregnants have limited physiological reserves and cardiovascular co- morbidities when compared to non-obese pregnant women. Spinal anaesthesia is the anaesthetic technique of choice for caesarean section. The haemodynamic changes associated with spinal anaesthesia pose the greatest hazard to the mother and the foetus and are exaggerated in obese pregnant women. However differences in the changes in haemodynamic variables such as cardiac output (CO), stroke volume (SV) and systemic vascular resistance (SVR) between obese and non-obese pregnant women having caesarean section (CS) under spinal anaesthesia have not been studied before. This study compares the haemodynamic changes after spinal anaesthesia for CS in non-obese and obese parturients in a single centre, prospective case control study, using LiDCOrapidV2. This LiDCOrapidV2 device is a noninvasive method of measuring haemodynamic variables. It is a single centre, prospective, case control study. The primary outcome compares the differences and variability in CO, SV and SVR between obese and non-obese parturients. The secondary outcomes include comparison of the correlation between changes in blood pressure (BP) and CO in each patient and the difference in BP between conventional intermittent oscillometric device and continuous LiDCORapidV2in each patient with a view to assess the need for measurement of cardiac output in obstetric anaesthesia

DETAILED DESCRIPTION:
Pregnancy is a state of physiological alteration as a result of increased oxygen demand and involves significant haemodynamic changes including sustained rises in cardiac output (CO) (by up to 30- 60%) and stroke volume (SV) (up to 30%) by virtue of increase in the blood volume This is associated with decrease in the systemic vascular resistance (SVR) and enhanced myocardial performance. When pregnancy is associated with obesity the cardiovascular system is further stressed. Obese pregnant women with a body mass index (BMI) more than 35kg/m2 pose significant health issue and are at risk for anaesthesia related maternal mortality. Several cases of sudden cardiac arrests of unexplained cause in obese pregnants have been reported. Obesity induced pathological changes have profound effects on cardiac endothelial and vascular function. Thus in pregnancy, obesity leads to further increase in blood volume and cardiac output proportionate to the amount of fat thus causing further volume overload of the heart. A study conducted with transthoracic echo showed a mean increase of around 550mls in cardiac output between obese and non-obese parturients in the third trimester. In contrast to the decrease in SVR that occurs in normal pregnancy, obesity by itself is associated with increased SVR by virtue of the increased sympathetic activity due to the effects of hormones including leptin, insulin and inflammatory mediators. This causes an increase in afterload 6, 8 thus offsetting the advantage of reduced afterload of normal pregnancy affecting the CO further. This combination of volume and pressure overload leads to systolic dysfunction. Furthermore the increase in heart rate of pregnancy in line with elevated cardiac output will decrease the diastolic interval and time for myocardial perfusion causing diastolic dysfunction. Thus obese pregnant patients may present with a systolic, diastolic or both systolic and diastolic dysfunction of the left ventricle. Associated obstructive sleep apneoa (OSA) and pulmonary hypertension may lead to right ventricular failure. These changes are further compromised in the third trimester due to aortocaval compression thus reducing cardiac output and placental perfusion. The large abdominal panniculus in obesity will further add to the uterine and vascular compression. It is thus evident that obese parturient women pose an increase in risk for cardiovascular compromise. As obesity is considered a global health care problem especially in women, anaesthetists are increasingly faced with the care of this high risk group of patients.9However there is paucity of evidence to quantify this cardiovascular compromise on obese pregnant women and guide provision of best care.

Regional anaesthesia has been the preferred technique of anaesthesia, especially in obese pregnant patients. Induction of spinal anaesthesia will cause profound haemodynamic changes that represent the greatest hazard to the mother and the foetus. Evidence suggests these haemodynamic changes are common after spinal anaesthesia and results in hypotension causing unconsciousness, maternal nausea and vomiting, dizziness including deleterious effects on the foetus like neonatal acidaemia and lower APGAR score. However because of the changes in peripheral vascular resistance, changes in maternal arterial pressure do not necessarily reflect changes in maternal cardiac output. These changes in cardiac output and associated oxygen delivery pose the greatest risk to the foetus.

A recent review of cardiovascular alterations in the parturient undergoing caesarean delivery with neuraxial anaesthesia showed that induction of spinal anaesthesia will lead to decrease in CO by 10-35% as measured by various invasive techniques. Although the patho-physiology of pregnancy and obesity and echocardiography findings gives us an understanding that these patients are more prone for severe hypotension and cardiovascular compromise the extent of alteration of haemodynamic variables in obese pregnant patients during spinal anaesthesia has not been studied previously. Our primary aim therefore is to investigate the haemodynamic alterations in obese parturient during spinal anaesthesia and compare it with those in non-obese parturient.

Traditionally clinicians and researchers have used heart rate (HR)and BP as surrogate markers of cardiac output during spinal anaesthesia. Managing maternal BP was considered as safe optimization of foetal wellbeing. Recent publications have emphasized that keeping BP at baseline is not an optimal strategy and maintaining CO is superior in maintaining uterine blood flow. In addition the correlation of the foetal compromise in the form of umbilical artery pH and umbilical artery pulsatality index was better related to SV and CO than BP and heart rate. 19 Thus measurement of CO is considered a better approach than BP in optimising oxygen delivery to the foetus.

Although pulmonary artery catheterization is a gold standard for measuring cardiac output it is not desirable to use routinely because of its invasiveness, patient compliance and its potential complications. Minimally invasive CO monitors like LiDCO plus has been validated and successfully used for this purpose, but still require an arterial line and is complex for routine use.

LiDCOrapidV2(LiDCO Group plc, LiDCO Limited, United Kingdom), incorporates the CNAPTM (continuous noninvasive arterial pressure) module that derives CO, SV, and SVR from a continuous noninvasive arterial waveform and analysed by the PulseCOTM algorithm avoiding invasive blood pressure measurements. This study studies the clinical application of the LIDCOrapidV2 and compares the haemodynamic variables in obese and non-obese pregnant women having CS under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients with BMI of less than 30 undergoing elective CS.
2. Obese pregnant patients with BMI of more than 35 undergoing elective CS

Exclusion Criteria:

1. Patients with other comorbidities like pre-eclampsia, eclampsia, essential hypertension, respiratory disease and compromised renal function.
2. Patients on long-term medication.
3. Patients having CS under epidural.
4. Patients having general anaesthesia.
5. Patients on antihypertensive medication.
6. Patients with BMI of 31-34.
7. Patients less than 36 weeks of gestation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Difference in the variation of cardiac output (CO) from baseline values between obese and non-obese parturients after spinal anaesthesia. | 18 months
  The change in cardiac output from baseline measured as milliliters/minute at predetermined intervals after spinal anaesthesia will be recorded in each group. The mean value of this change in each group will be compared for each recording and the difference in the change between the two groups will be reported.

SECONDARY OUTCOMES:
Mean difference in the amount of vasopressors infused in millilitres/hour between non-obese and obese pregnant women. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Kumar, FRCA, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Maternity Hospital, Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No